CLINICAL TRIAL: NCT00534196
Title: Japanese Prostate Cancer Outcome Study by Permanent I-125 Seed Implantation [J-POPS]
Brief Title: Implant Radiation Therapy Using Radioactive Iodine in Treating Patients With Localized Prostate Cancer
Acronym: J-POPS
Status: Completed | Type: Observational
Sponsor: Translational Research Center for Medical Innovation, Kobe, Hyogo, Japan (Other)
Collaborators: Kurosawa Hospital (Unknown)
Responsible Party: Sponsor
Other Study IDs: CDR0000562726; TUSM-BRI-GU-04-01
Record Dates: First submitted 2007-09-20; First posted 2007-09-24 (Estimated); Last update posted 2023-06-26 (Actual); Status verified 2022-05

CONDITIONS: Prostate Cancer
Keywords: recurrent prostate cancer; stage I prostate cancer; stage IIB prostate cancer; stage IIA prostate cancer; stage III prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Brachytherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Group under operation of brachytherapy: Patients with histologically confirmed adenocarcinoma of the prostate and who are planning to undergo brachytherapy with PI (permanent iodine) or combination of PI with other tratement.
  Interventions: Radiation: Permanent iodine-125 (Brachytherapy)

INTERVENTIONS:
Radiation: Permanent iodine-125 (Brachytherapy) — Observational research was conducted by grouping Brachytherapy with/without PI (permanent iodine) seed implantation.

SUMMARY:
RATIONALE: Implant radiation therapy delivers a high dose of radiation directly to the tumor may kill more tumor cells and cause less damage to normal tissue.

PURPOSE: This clinical trial is studying the side effects and how well implant radiation therapy using radioactive iodine works in treating patients with localized prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* To determine the efficacy of permanent brachytherapy with iodine I 125 seeds in patients with localized prostate cancer.
* To determine the safety of this therapy in these patients.

OUTLINE: This is a multicenter study.

Patients undergo permanent brachytherapy seed implantation comprised of iodine I 125 into the prostate. Some patients may receive combination treatment (e.g., external beam radiation therapy (EBRT) or hormone therapy in addition to brachytherapy).

Quality of life and the International Prostate Symptom Score (IPSS) is assessed and compared.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Clinically and histologically confirmed localized prostate cancer

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* No prior or concurrent surgery
* No prior or concurrent radiotherapy
* Prior chemotherapy, hormonal therapy, and biologic therapy allowed

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients in Japan who is histologically confirmed adenocarcinoma of the prostate and planning to undergo treatment with PI or combination of PI with other treatment.
Sampling Method: Non-Probability Sample
Enrollment: 6927 (Actual)
Dates: Start 2005-07; Primary Completion 2016-11-30 (Actual); Study Completion 2021-12-13 (Actual)

PRIMARY OUTCOMES:
PSA relapse-free survival | 5 years
  Defined as the duration from enrollment to the date of biological relapse, which was defined as three consecutive prostate specific antigen (PSA) rises in the reflex range of 1.0 ng/ml or greater, and the date of failure was the midpoint between the first day that showed PSA levels 1.0 ng/ml or greater and the last day in which the level was below 1.0 ng/ml.

SECONDARY OUTCOMES:
Progression free survival (PFS) | 5 years
  Dration from enrollment to the date of biochemical relapse or clinical relapse, overall survival (OS), cause-specific survival (CSS).
Quality of life | Baseline, Month 3, 12, 24 and 36
  The Japanese version of the SF-8 (the MOS 8 item Short-Form Health Survey), the Japanese version of the Extended Prostate Cancer Index Composite (EPIC) are used for characterizing Longitudinal changes in health-related quality of life (HRQOL), and the EPIC was used to investigate disease-specific quality of life (disease-specific QOL). Patients enrolled between July 2005 - June 2007 will be evaluated.
IPSS score | Baseline, Month 3, 12, 24 and 36
  Evaluated by International Prostate Syndrom Score (IPSS)
Adverse events | 36 months
  Types and severities of adverse events from date of starting protocol treatment until the first 30 months after date of finishing the treatment are evaluated in the most serious adverse events of each reporting period according to Japanese version of the National Cancer Institute Common Terminology Criteria for Adverse Events version 3.0 (CTCAE v3.0) by Translational Research Informatics Center.

CONTACTS AND LOCATIONS:
Overall Officials: Shiro Saito, MD, PhD, Study Chair — National Hospital Organization Tokyo Medical Center
Locations (31):
- Japan (31):
  - Fujita Health University, Toyoake, Aichi-ken
  - Shikoku Cancer Center, Matsuyama, Ehime
  - Ehime University Hospital, Tōon, Ehime
  - Isesaki Municipal Hospital, Isesaki, Gunma
  - Gunma University Graduate School of Medicine, Maebashi, Gunma
  - Kurosawa Hospital, Takasaki, Gunma
  - Sapporo Medical University, Sapporo, Hokkaido
  - Translational Research Informatics Center, Kobe, Hyōgo
  - Ibaraki Prefectural Central Hospital, Kasama, Ibaraki
  - Kagawa University Hospital, Hiragi, Kagawa-ken
  - Osaka University Graduate School of Medicine, Suita, Osaka
  - National Hospital Organization - Saitama National Hospital, Wako, Saitama
  - Shiga University of Medical Science, Ōtsu, Shiga
  - Shimane University Hospital, Izumo, Shimane
  - University of Fukui Hospital, Fukui
  - Hamanomachi Hospital, Fukuoka
  - Kyushu University Hospital, Fukuoka
  - Gifu University Graduate School of Medicine, Gifu
  - Gunma Cancer Center, Gunma
  - Kitasato University School of Medicine, Kanagawa
  - Kyoto Prefectural University of Medicine, Kyoto
  - Nagasaki University Hospital, Nagasaki
  - Okayama University Medical School, Okayama
  - Saitama Cancer Center, Saitama
  - Tokushima University Hospital, Tokushima
  - Nippon Medical School, Tokyo
  - University of Tokyo Hospital, Tokyo
  - Cancer Institute Hospital of Japanese Foundation for Cancer Research, Tokyo
  - National Hospital Organization - Tokyo Medical Center, Tokyo
  - Keio University School of Medicine, Tokyo
  - Tokyo Women's Medical University, Tokyo

REFERENCES:
- [Derived] Ito K, Saito S, Yorozu A, Kojima S, Kikuchi T, Higashide S, Aoki M, Koga H, Satoh T, Ohashi T, Nakamura K, Katayama N, Tanaka N, Nakano M, Shigematsu N, Dokiya T, Fukushima M; J-POPS Investigators. Nationwide Japanese Prostate Cancer Outcome Study of Permanent Iodine-125 Seed Implantation (J-POPS): first analysis on survival. Int J Clin Oncol. 2018 Dec;23(6):1148-1159. doi: 10.1007/s10147-018-1309-0. Epub 2018 Jun 22. PMID 29934842
- [Derived] Nakano M, Yorozu A, Saito S, Sugawara A, Maruo S, Kojima S, Kikuchi T, Fukushima M, Dokiya T, Yamanaka H. Seed migration after transperineal interstitial prostate brachytherapy by using loose seeds: Japanese prostate cancer outcome study of permanent iodine-125 seed implantation (J-POPS) multi-institutional cohort study. Radiat Oncol. 2015 Nov 14;10:228. doi: 10.1186/s13014-015-0532-3. PMID 26577301
- [Derived] Saito S, Ito K, Yorozu A, Aoki M, Koga H, Satoh T, Ohashi T, Shigematsu N, Maruo S, Kikuchi T, Kojima S, Dokiya T, Fukushima M, Yamanaka H. Nationwide Japanese Prostate Cancer Outcome Study of Permanent Iodine-125 Seed Implantation (J-POPS). Int J Clin Oncol. 2015 Apr;20(2):375-85. doi: 10.1007/s10147-014-0704-4. Epub 2014 May 21. PMID 24840041